CLINICAL TRIAL: NCT04640441
Title: Effect of Sit-to-Stand Intervention in the Intensive Care Unit Survivors: A Randomized Controlled Trial
Brief Title: Effect of Sit-to-Stand Intervention in the Intensive Care Unit Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202007109RINB
Record Dates: First submitted 2020-09-10; First posted 2020-11-23 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-01

CONDITIONS: Unable to Sit-to-stand; ICU Survivor
Keywords: Sit-to-stand; Functional decline; Intensive care units; Nursing intervention; Randomized controlled trial

STUDY DESIGN:
Intervention Model Description: Participants who were screened as failure to sit-to-stand after discharged from medication ICU 48 hours were enrolled in the study. In the assignment procedure, participants were stratified by "able to remain sitting upright without falling" or "unable to remain sitting upright" and then 1:1 randomly assigned to the intervention or usual care groups. Participants in intervention group received both usual care and an STS care once daily for two weeks or discharged within two weeks or death. In contrast, control group will accept regular care. Participants were followed for one year after ICU discharge at 5 point:48 hours, 14day, 1, 3, and 12 months. A comprehensive functional evaluation (success rate of sit-to-stand, scores of FSS-ICU, scores of MRC scale, muscle strength at knee extensors, scores of barthel index for ADL, scores of IADL, walking distance by 6-minute walk test, numbers of sit-to-stand repetitions in 30 seconds) and rates of bed-bound status and mortality were performed.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Participants in the control group received usual care.
- Sit-to-stand care group (Experimental): Intervention was provided once daily by trained nurses for a maximum of 14 days or until hospital discharge or death.
  Interventions: Other: Sit-to-stand care

INTERVENTIONS:
Other: Sit-to-stand care — 1. Passive range of motion(ROM) exercise of lower legs, active ROM exercise of lower legs, and sitting balance exercise, 20~30 min, once daily.
  2. Anti-gravity ROM exercise of lower leg, resistance exercise of low leg, and sitting balance exercise, 20~30min, once daily.
  3. Stepping exercise and sit-to-stand exercise, 20~30min, once daily.
  Arms: Sit-to-stand care group

SUMMARY:
"Sit-to-stand" is key to independent living. For intensive care unit (ICU) survivors, failure to perform sit-to-stand results in bed-bound status, unable participating in important activities of daily living (ADLs) or instrumental ADLs. Recent studies indicated that 31% of ICU survivors remained bed-bound and unable to "sit-to-stand" after returning home. Our preliminary findings further indicated that 70% of ICU survivors who had the ICU-acquired weakness (ICU-AW) were unable to "sit-to-stand" one-month after ICU discharge.

The aim of this 3-year research project was to develop a feasible and effective "sit-to-stand" care (STS Care). A randomized controlled trial (RCT) design is proposed to examine effects of the STS Care in improving ICU patients' "sit-to-stand" ability, physical function, and rates of bed-bound and mortality one year following ICU discharge.

The trial was approved by the Human Research Ethics Committee at the study site before enrollment. Adult ICU patients (≥ 20 years) admitted consecutively to six medical ICUs of a university affiliated medical center was eligible for the study if they were unable to "sit-to-stand" independently at ICU discharge. Upon signing informed consent, participants will be first stratified by "able to remain sitting upright without falling" or "unable to remain sitting upright" and then randomized separately into the intervention or usual care groups, according to computer-generated randomization tables. Participants in the intervention group received both usual care and the STS Care.

The hospital-based (up to 14 days) STS Care, which was provided daily by the same trained nurse, consisted of nurse-supervised anti-gravity and resistant exercise (intensity based on patients' tolerance), repetitive sit-to-stand practice, and advice on sit-to-stand strategies. A comprehensive functional evaluation (success rate of sit to stand, scores of FSS-ICU, scores of MRC muscle scale, muscle strength at knee extensors, scores of the barthel index for activities of daily living (ADL), scores of instrumental activities of daily living scale (IADL), the walking distance by the 6-minute walk test, numbers of sit-to-stand repetitions in 30 seconds, rate of bed-bound status, rate of mortality) was assessed by blinded research nurses after ICU discharge at 5 time points:48hours, 14 day, 1, 3, and 12 months.

DETAILED DESCRIPTION:
For this stratified randomization and single blinding study, participants (≧20 years) who are screened with failed sit-to-stand ability after discharged from the National Taiwan University Hospital medication ICU 48hours will be enrolled in the study. In the assignment procedure, the participants will be stratified by a stabilized sitting posture and unable stabilized sitting posture, and then the participants are randomized to the experiment group and control group. The experiment group will accept regular care and an extra STS bedside care protocol once a day for two weeks or discharged within two weeks. In contrast, the control group will accept regular care.

All participants will be followed for one year after ICU discharge at 5 time points:48 hours, 14day,1, 3, 12 months. A comprehensive functional evaluation (success rate of sit to stand, scores of FSS-ICU, scores of MRC muscle scale, muscle strength at knee extensors, scores of the barthel index for activities of daily living (ADL), scores of instrumental activities of daily living scale (IADL), the walking distance by the 6-minute walk test, numbers of sit-to-stand repetitions in 30 seconds, rate of bed-bound status, rate of mortality) will be performed. Estimated 206 participants will be enrolled and followed one year after ICU discharge.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 years or older.
* Admitted for ICU treatment > 2 days.
* Unable to sit-to-stand by ICU discharge.

Exclusion Criteria:

* Unable to follow command.
* Bedridden before index hospitalization.
* Ventilator dependent after ICU discharge .
* Received palliative care.
* Co-morbidities of the trunk or lower limbs unable to ambulate due to neuromuscular or musculoskeletal etiology (e.g. CVA, spinal cord injury, amputation or fracture of lower limb).
* Placed on droplet or contact precausion (e.g. Open TB, SARS, COVID-19 )

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-11-08 (Actual)

PRIMARY OUTCOMES:
Sit-to-stand independently (percent) | Baseline within 48 hours. 14 day, 1, and 3 months after ICU discharge.
  Evaluated by one successful and independent sit-to-stand, allowed armrest use
scores of FSS-ICU | Baseline within 48 hours. 14 day, 1, and 3 months after ICU discharge.
  The FSS-ICU use 7-points score to evaluated 5 functional tasks, which includes rolling, supine-to -sit transfer, unsupported sitting, sit-to-stand transfer, and ambulation. Score range from 0 to 35, higher score indicated better physical performance.
scores of MRC muscle scale | Baseline within 48 hours. 1, 3, and 12 months after ICU discharge.
  Measured by medical research council scale (MRC) in score, range from 0 to 60 score, higher score indicated better muscle strength
muscle strength(kg) at knee extensors | Baseline within 48 hours. 14 day, 1, 3, and 12 months after ICU discharge.
  Measured by Hoggan MicroFET®2 in kg
30-second sit-to-stand test | 14day, 1, and 3 months after ICU discharge.
  Measured by recording the numbers of sit-to-stand a person can complete in 30 seconds

SECONDARY OUTCOMES:
Barthel index for activities of daily living (ADL) | Baseline within 48 hours. 1, 3, and 12 months after ICU discharge.
  Measured by ADL in score, range from 0-100 score, higher score indicated health condition
Instrumental activities of daily living scale (IADL) | Baseline within 48 hours. 1, 3, and 12 months after ICU discharge.
  Measured by IADL in score, range from 0 to 8 score, higher score indicated better health condition
Rate of bed-bound status (percent) | 1, 3, and 12 months after ICU discharge.
  Obtained by family interview and medical record
Rate of mortality (percent) | 1, 3, and 12 months after ICU discharge.
  Obtained by family interview and medical record
The 6 minute walk test | 3 and 12 months after ICU discharge.
  Measured by walked distance in 6 minutes(6MWT) in meter, range from 400 to 700 meters, higher value indicated better global health condition

CONTACTS AND LOCATIONS:
Locations (1):
- Cheryl, Chia-Hui Chen, PhD, Taipei, National Taiwan University Hospital, Taiwan

REFERENCES:
- [Background] Applebaum EV, Breton D, Feng ZW, Ta AT, Walsh K, Chasse K, Robbins SM. Modified 30-second Sit to Stand test predicts falls in a cohort of institutionalized older veterans. PLoS One. 2017 May 2;12(5):e0176946. doi: 10.1371/journal.pone.0176946. eCollection 2017. PMID 28464024
- [Background] Bednarik J, Vondracek P, Dusek L, Moravcova E, Cundrle I. Risk factors for critical illness polyneuromyopathy. J Neurol. 2005 Mar;252(3):343-51. doi: 10.1007/s00415-005-0654-x. Epub 2005 Mar 30. PMID 15791390
- [Background] Bloomfield SA. Changes in musculoskeletal structure and function with prolonged bed rest. Med Sci Sports Exerc. 1997 Feb;29(2):197-206. doi: 10.1097/00005768-199702000-00006. PMID 9044223
- [Background] Bodilsen AC, Klausen HH, Petersen J, Beyer N, Andersen O, Jorgensen LM, Juul-Larsen HG, Bandholm T. Prediction of Mobility Limitations after Hospitalization in Older Medical Patients by Simple Measures of Physical Performance Obtained at Admission to the Emergency Department. PLoS One. 2016 May 19;11(5):e0154350. doi: 10.1371/journal.pone.0154350. eCollection 2016. PMID 27195499
- [Background] Bohannon RW, Bubela DJ, Wang YC, Magasi SR, Gershon RC. Adequacy of belt-stabilized testing of knee extension strength. J Strength Cond Res. 2011 Jul;25(7):1963-7. doi: 10.1519/JSC.0b013e3181e4f5ce. PMID 21399535
- [Background] Bruun IH, Maribo T, Norgaard B, Schiottz-Christensen B, Mogensen CB. A prediction model to identify hospitalised, older adults with reduced physical performance. BMC Geriatr. 2017 Dec 7;17(1):281. doi: 10.1186/s12877-017-0671-5. PMID 29216838
- [Background] Ciesla N, Dinglas V, Fan E, Kho M, Kuramoto J, Needham D. Manual muscle testing: a method of measuring extremity muscle strength applied to critically ill patients. J Vis Exp. 2011 Apr 12;(50):2632. doi: 10.3791/2632. PMID 21505416
- [Background] Connolly B, Thompson A, Douiri A, Moxham J, Hart N. Exercise-based rehabilitation after hospital discharge for survivors of critical illness with intensive care unit-acquired weakness: A pilot feasibility trial. J Crit Care. 2015 Jun;30(3):589-98. doi: 10.1016/j.jcrc.2015.02.002. Epub 2015 Feb 7. PMID 25703957
- [Background] De Jonghe B, Sharshar T, Lefaucheur JP, Authier FJ, Durand-Zaleski I, Boussarsar M, Cerf C, Renaud E, Mesrati F, Carlet J, Raphael JC, Outin H, Bastuji-Garin S; Groupe de Reflexion et d'Etude des Neuromyopathies en Reanimation. Paresis acquired in the intensive care unit: a prospective multicenter study. JAMA. 2002 Dec 11;288(22):2859-67. doi: 10.1001/jama.288.22.2859. PMID 12472328
- [Background] Fan E, Dowdy DW, Colantuoni E, Mendez-Tellez PA, Sevransky JE, Shanholtz C, Himmelfarb CR, Desai SV, Ciesla N, Herridge MS, Pronovost PJ, Needham DM. Physical complications in acute lung injury survivors: a two-year longitudinal prospective study. Crit Care Med. 2014 Apr;42(4):849-59. doi: 10.1097/CCM.0000000000000040. PMID 24247473
- [Background] Fetterplace K, Beach LJ, MacIsaac C, Presneill J, Edbrooke L, Parry SM, Rechnitzer T, Curtis R, Berney S, Deane AM, Denehy L. Associations between nutritional energy delivery, bioimpedance spectroscopy and functional outcomes in survivors of critical illness. J Hum Nutr Diet. 2019 Dec;32(6):702-712. doi: 10.1111/jhn.12659. Epub 2019 Apr 29. PMID 31034122
- [Background] Fortes-Filho SQ, Aliberti MJR, Apolinario D, Melo-Fortes JA, Sitta MC, Jacob-Filho W, Garcez-Leme LE. Role of Gait Speed, Strength, and Balance in Predicting Adverse Outcomes of Acutely Ill Older Outpatients. J Nutr Health Aging. 2020;24(1):113-118. doi: 10.1007/s12603-019-1279-6. PMID 31886817
- [Background] Gross MM, Stevenson PJ, Charette SL, Pyka G, Marcus R. Effect of muscle strength and movement speed on the biomechanics of rising from a chair in healthy elderly and young women. Gait Posture. 1998 Dec 1;8(3):175-185. doi: 10.1016/s0966-6362(98)00033-2. PMID 10200407
- [Background] Huang M, Chan KS, Zanni JM, Parry SM, Neto SG, Neto JA, da Silva VZ, Kho ME, Needham DM. Functional Status Score for the ICU: An International Clinimetric Analysis of Validity, Responsiveness, and Minimal Important Difference. Crit Care Med. 2016 Dec;44(12):e1155-e1164. doi: 10.1097/CCM.0000000000001949. PMID 27488220
- [Background] Iwashyna TJ, Ely EW, Smith DM, Langa KM. Long-term cognitive impairment and functional disability among survivors of severe sepsis. JAMA. 2010 Oct 27;304(16):1787-94. doi: 10.1001/jama.2010.1553. PMID 20978258
- [Background] Kaukonen KM, Bailey M, Suzuki S, Pilcher D, Bellomo R. Mortality related to severe sepsis and septic shock among critically ill patients in Australia and New Zealand, 2000-2012. JAMA. 2014 Apr 2;311(13):1308-16. doi: 10.1001/jama.2014.2637. PMID 24638143
- [Background] Kiriella JB, Araujo T, Vergara M, Lopez-Hernandez L, Cameron JI, Herridge M, Gage WH, Mathur S. Quantitative Evaluation of Muscle Function, Gait, and Postural Control in People Experiencing Critical Illness After Discharge From the Intensive Care Unit. Phys Ther. 2018 Jan 1;98(1):8-15. doi: 10.1093/ptj/pzx102. PMID 29088390
- [Background] Ko RE, Lee H, Jung JH, Lee HO, Sohn I, Yoo H, Ko JY, Suh GY, Chung CR. Simple functional assessment at hospital discharge can predict long-term outcomes of ICU survivors. PLoS One. 2019 Apr 4;14(4):e0214602. doi: 10.1371/journal.pone.0214602. eCollection 2019. PMID 30947283
- [Background] Kress JP, Hall JB. ICU-acquired weakness and recovery from critical illness. N Engl J Med. 2014 Jul 17;371(3):287-8. doi: 10.1056/NEJMc1406274. No abstract available. PMID 25014703
- [Background] Lawton MP, Brody EM. Assessment of older people: self-maintaining and instrumental activities of daily living. Gerontologist. 1969 Autumn;9(3):179-86. No abstract available. PMID 5349366
- [Background] LeBlanc AD, Schneider VS, Evans HJ, Pientok C, Rowe R, Spector E. Regional changes in muscle mass following 17 weeks of bed rest. J Appl Physiol (1985). 1992 Nov;73(5):2172-8. doi: 10.1152/jappl.1992.73.5.2172. PMID 1474100
- [Background] Martins J, da Silva JR, da Silva MRB, Bevilaqua-Grossi D. Reliability and Validity of the Belt-Stabilized Handheld Dynamometer in Hip- and Knee-Strength Tests. J Athl Train. 2017 Sep;52(9):809-819. doi: 10.4085/1062-6050-52.6.04. Epub 2017 Aug 8. PMID 28787180
- [Background] Matsufuji S, Shoji T, Yano Y, Tsujimoto Y, Kishimoto H, Tabata T, Emoto M, Inaba M. Effect of chair stand exercise on activity of daily living: a randomized controlled trial in hemodialysis patients. J Ren Nutr. 2015 Jan;25(1):17-24. doi: 10.1053/j.jrn.2014.06.010. Epub 2014 Sep 4. PMID 25194621
- [Background] McAllister LS, Palombaro KM. Modified 30-Second Sit-to-Stand Test: Reliability and Validity in Older Adults Unable to Complete Traditional Sit-to-Stand Testing. J Geriatr Phys Ther. 2020 Jul/Sep;43(3):153-158. doi: 10.1519/JPT.0000000000000227. PMID 30807554
- [Background] Puthucheary ZA, Rawal J, McPhail M, Connolly B, Ratnayake G, Chan P, Hopkinson NS, Phadke R, Dew T, Sidhu PS, Velloso C, Seymour J, Agley CC, Selby A, Limb M, Edwards LM, Smith K, Rowlerson A, Rennie MJ, Moxham J, Harridge SD, Hart N, Montgomery HE. Acute skeletal muscle wasting in critical illness. JAMA. 2013 Oct 16;310(15):1591-600. doi: 10.1001/jama.2013.278481. PMID 24108501
- [Background] Ragavan, V. K., Greenwood, K. C., & Bibi, K. (2016). The Functional Status Score for the Intensive Care Unit Scale: is it reliable in the intensive care unit? Can it be used to determine discharge placement? Journal of Acute Care Physical Therapy, 7(3), 93-100.
- [Background] Reychler G, Boucard E, Peran L, Pichon R, Le Ber-Moy C, Ouksel H, Liistro G, Chambellan A, Beaumont M. One minute sit-to-stand test is an alternative to 6MWT to measure functional exercise performance in COPD patients. Clin Respir J. 2018 Mar;12(3):1247-1256. doi: 10.1111/crj.12658. Epub 2017 Jun 15. PMID 28621019
- [Background] Richtrmoc, M. K., Leite, W. S., Barros, C. E. S. R., Lima, A. M. S., Azevedo, A. M., Vasconcelos, A. P., . . . Campos, S. L. (2017). Admission status of respiratory, peripheral muscle strengths deficits and functionality in non-ventilated patients under intensive care. European Respiratory Journal, 50(suppl 61), PA2111. doi:10.1183/1393003.congress-2017.PA2111
- [Background] Ridley EJ, Parke RL, Davies AR, Bailey M, Hodgson C, Deane AM, McGuinness S, Cooper DJ. What Happens to Nutrition Intake in the Post-Intensive Care Unit Hospitalization Period? An Observational Cohort Study in Critically Ill Adults. JPEN J Parenter Enteral Nutr. 2019 Jan;43(1):88-95. doi: 10.1002/jpen.1196. Epub 2018 Jun 20. PMID 29924393
- [Background] Rikli RE, Jones CJ. Development and validation of criterion-referenced clinically relevant fitness standards for maintaining physical independence in later years. Gerontologist. 2013 Apr;53(2):255-67. doi: 10.1093/geront/gns071. Epub 2012 May 20. PMID 22613940
- [Background] Riley PO, Krebs DE, Popat RA. Biomechanical analysis of failed sit-to-stand. IEEE Trans Rehabil Eng. 1997 Dec;5(4):353-9. doi: 10.1109/86.650289. PMID 9422460
- [Background] Roebroeck ME, Doorenbosch CA, Harlaar J, Jacobs R, Lankhorst GJ. Biomechanics and muscular activity during sit-to-stand transfer. Clin Biomech (Bristol). 1994 Jul;9(4):235-44. doi: 10.1016/0268-0033(94)90004-3. PMID 23916233
- [Background] Sacanella E, Perez-Castejon JM, Nicolas JM, Masanes F, Navarro M, Castro P, Lopez-Soto A. Functional status and quality of life 12 months after discharge from a medical ICU in healthy elderly patients: a prospective observational study. Crit Care. 2011;15(2):R105. doi: 10.1186/cc10121. Epub 2011 Mar 28. PMID 21443796
- [Background] Sainsbury A, Seebass G, Bansal A, Young JB. Reliability of the Barthel Index when used with older people. Age Ageing. 2005 May;34(3):228-32. doi: 10.1093/ageing/afi063. PMID 15863408
- [Background] Schenkman M, Berger RA, Riley PO, Mann RW, Hodge WA. Whole-body movements during rising to standing from sitting. Phys Ther. 1990 Oct;70(10):638-48; discussion 648-51. doi: 10.1093/ptj/70.10.638. PMID 2217543
- [Background] Shah S, Vanclay F, Cooper B. Improving the sensitivity of the Barthel Index for stroke rehabilitation. J Clin Epidemiol. 1989;42(8):703-9. doi: 10.1016/0895-4356(89)90065-6. PMID 2760661
- [Background] Slaughter SE, Wagg AS, Jones CA, Schopflocher D, Ickert C, Bampton E, Jantz A, Milke D, Schalm C, Lycar C, Estabrooks CA. Mobility of Vulnerable Elders study: effect of the sit-to-stand activity on mobility, function, and quality of life. J Am Med Dir Assoc. 2015 Feb;16(2):138-43. doi: 10.1016/j.jamda.2014.07.020. Epub 2014 Sep 27. PMID 25271194
- [Background] Strassmann A, Steurer-Stey C, Lana KD, Zoller M, Turk AJ, Suter P, Puhan MA. Population-based reference values for the 1-min sit-to-stand test. Int J Public Health. 2013 Dec;58(6):949-53. doi: 10.1007/s00038-013-0504-z. Epub 2013 Aug 24. PMID 23974352
- [Background] Thomas S, Burridge JH, Pohl M, Oehmichen F, Mehrholz J. Recovery of sit-to-stand function in patients with intensive-care-unit-acquired muscle weakness: Results from the General Weakness Syndrome Therapy cohort study. J Rehabil Med. 2016 Oct 12;48(9):793-798. doi: 10.2340/16501977-2135. PMID 27670853
- [Background] Thrush A, Rozek M, Dekerlegand JL. The clinical utility of the functional status score for the intensive care unit (FSS-ICU) at a long-term acute care hospital: a prospective cohort study. Phys Ther. 2012 Dec;92(12):1536-45. doi: 10.2522/ptj.20110412. Epub 2012 Sep 6. PMID 22956427
- [Background] Vaidya T, Chambellan A, de Bisschop C. Sit-to-stand tests for COPD: A literature review. Respir Med. 2017 Jul;128:70-77. doi: 10.1016/j.rmed.2017.05.003. Epub 2017 May 15. PMID 28610673
- [Background] van der Schaaf M, Dettling DS, Beelen A, Lucas C, Dongelmans DA, Nollet F. Poor functional status immediately after discharge from an intensive care unit. Disabil Rehabil. 2008;30(23):1812-8. doi: 10.1080/09638280701673559. PMID 19031208
- [Background] van Zanten ARH, De Waele E, Wischmeyer PE. Nutrition therapy and critical illness: practical guidance for the ICU, post-ICU, and long-term convalescence phases. Crit Care. 2019 Nov 21;23(1):368. doi: 10.1186/s13054-019-2657-5. PMID 31752979
- [Background] Waters A, Hill K, Jenkins S, Johnston C, Mackney J. Discordance Between Distance Ambulated as Part of Usual Care and Functional Exercise Capacity in Survivors of Critical Illness Upon Intensive Care Discharge: Observational Study. Phys Ther. 2015 Sep;95(9):1254-63. doi: 10.2522/ptj.20140282. Epub 2015 Apr 2. PMID 25838336